CLINICAL TRIAL: NCT02499354
Title: Double-blind Comparator of Efficacy of Oral (Ferrous Sulfate) vs. Intravenous Iron (Ferumoxytol) for Treatment of the Restless Legs Syndrome (RLS) Occurring With Iron Deficient Anemia (IDA)
Brief Title: Pilot Study: Randomized, Placebo-controlled Comparator Trial of IV vs Oral Iron Treatment of RLS With IDA. (IVOR-IDA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Auerbach Hematology Oncology Associates P C (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Auerbach MD, Dr. Michael Auerbach, Auerbach Hematology Oncology Associates P C
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IVOR-IDA
Record Dates: First submitted 2015-07-13; First posted 2015-07-16 (Estimated); Results first posted 2023-08-15 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Restless Legs Syndrome; Iron Deficiency Anemia
MeSH Terms: conditions — Restless Legs Syndrome; Anemia, Iron-Deficiency | interventions — ferryl iron; ferrous sulfate; Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Iron (Active Comparator): Ferrous Sulfate 325mg (oral) tabs morning and evening
  Interventions: Drug: Ferrous sulfate
- IV Iron (Active Comparator): Ferumoxytol intravenous (IV) 1020 mg - 2 vials of 510 mg (IV push, 2-3 mins) each given 2-7 days apart
  Interventions: Drug: Ferumoxytol intravenous

INTERVENTIONS:
Drug: Ferumoxytol intravenous — IV iron, 2 vials of 510 mg given 2-7 days apart
  Other Names: IV iron
  Arms: IV Iron
Drug: Ferrous sulfate — Oral iron, 325 mg tabs taken morning and evening
  Other Names: Oral iron
  Arms: Oral Iron

SUMMARY:
The purpose of the study is to determine the relative effect size of standard IV and oral iron treatment of RLS with Iron deficiency anemia (IDA) and to determine the time course of treatment response.

DETAILED DESCRIPTION:
The restless legs syndrome (RLS) (also known as Willis Ekbom Disease) occurs in about 1/3rd of patients with iron deficiency anemia (IDA). Treatment correcting the IDA is expected to also be effective for reducing or eliminating the RLS with IDA. Two accepted treatments for IDA (oral ferrous sulfate, intravenous ferumoxytol) will be compared for efficacy and speed to response for treatment of RLS occurring with IDA (RLS-IDA). In this study 70 RLS-IDA patients will be randomly assigned 35 each to oral or IV iron treatment using double-blind procedures. Primary outcome with be determined at 6 weeks of treatment with a follow-up at 12 months after treatment. Non-responders at 6 weeks after treatment may, if they qualify, have an open-label IV iron treatment and they will be followed with the same evaluations used after the first set of IV iron treatments.

Both oral and IV iron are considered standard treatments for IDA. These same treatments also reduce RLS symptoms. The treatment doses are those accepted for treatment of RLS and also appropriate for treatment for RLS-IDA. Choosing doses equivalent to those for the treatment of RLS without IDA will allow a comparison with that literature. The investigators will therefore use for oral iron ferrous sulfate 325mg taken twice a day matching the dose used in the study of oral iron treatment for RLS without anemia. For IV iron investigators will use ferumoxytol, provided by the sponsor, two doses of 510 mg spaced 2 to 7 days apart. This is the FDA approved dose for treatment of IDA with end stage renal disease.

The study is a randomized, comparative open label study to evaluate effect size and time course of treatment response for RLS-IDA over 6 weeks with a 46-week follow-up extension. Two medications and placebos will be used, as described above, with equal random assignment to both groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RLS based on questionnaire and confirmed by Hopkins telephone Diagnostic Interview conducted by investigators or clinicians part of the study.
* Iron deficiency anemia defined as ID either ferritin <20 mcg/l, Tsat <19%, anemia Hgb <13 for both males and females.
* Willingness to use contraceptive to avoid pregnancy: Women have to be surgically sterile, post-menopausal, or use one of the following contraceptives during the whole study period and after the study has ended for at least 5 times plasma biological half-life of the investigational medicinal product: intrauterine devices or hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices, or injections with prolonged release).
* Willingness to participate and signing the informed consent form.

Exclusion Criteria:

* Iron overload or disturbances in utilization of iron (e.g. haemochromatosis and haemosiderosis)
* Decompensated liver cirrhosis or active hepatitis (ALAT > 3 times upper limit of normal)
* Serum ferritin > 500 ng/mL or transferrin saturation >40%
* Active acute or chronic infections (assessed by clinical judgement that may be indicated by White Blood Cells (WBC) and C-Reactive Protein (CRP) when these are available)
* Rheumatoid arthritis with symptoms or signs of active inflammation
* Pregnant and nursing women
* History of multiple allergies
* Known hypersensitivity to parenteral or oral iron or any excipients in the drug products
* Previous IV iron treatment for RLS
* Other iron treatment or blood transfusion within 4 weeks prior to the screening or treatment visit
* Planned elective surgery during the study
* Current (past 4 weeks) use of drugs that treat RLS, e.g. opioids, alpha-2-delta anti-depressants, dopaminergics (dopamine promoters, dopamine antagonists/blockers)
* Any other medical condition that, in the opinion of Investigator, may cause the subject to be unsuitable for the completion og the study or place the subject at potential risk from being in the study, e.g. a malignancy, uncontrolled hypertension, unstable ischemic heart disease, or uncontrolled diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Auerbach, MD, Principal Investigator — Auerbach Hematology and Oncology Associates, PC
Locations (1):
- Auerbach Hematology Oncology Assoc, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Iron: Ferrous Sulfate 325mg (oral) tabs morning and evening
  Ferrous sulfate: Oral iron, 325 mg tabs taken morning and evening
  In this arm participants also received intravenous normal saline as part of a double blind, double dummy design
- IV Iron: Ferumoxytol intravenous (IV) 1020 mg - 2 vials of 510 mg (IV push, 2-3 mins) each given 2-7 days apart
  Ferumoxytol intravenous: IV iron, 2 vials of 510 mg given 2-7 days apart
  In this arm participants received oral vitamin C as part of a double blind, double dummy design
Period: Overall Study
Arm/Group | Oral Iron | IV Iron
Started | 46 | 47
Completed | 45 | 47
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Iron | IV Iron | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 44 | 45 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 40 | 84
  Male | 2 | 7 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 39 | 42 | 81
  Unknown or Not Reported | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 46 | 47 | 93

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Restless Legs Syndrome Rating Scale
Description: Change in International Restless Legs Severity Scale (IRLS) score reflecting RLS severity on the scale of 0-40. The higher the negative score the better the outcome
Time Frame: Baseline and at 6 weeks after treatment
Population: Those participants with baseline data and at 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Iron | IV Iron
Number analyzed (Participants) | 45 | 47
units on a scale | -14.0000 (9.75) | -9.7353 (8.33)
Statistical Analysis 1: Comparison: Oral Iron vs IV Iron; Test type: Superiority; p = 0.2742, t-test, 1 sided

2. Primary Outcome: Percentage of Participants With Improvement on Clinical Global Impression Scale
Description: Seven questions ranging from Very Much Improved to Very Much Worse: Participant had to be at least Very Much Improved to be considered as having improved. The CGI scale consisted of one question.
Time Frame: Six weeks
Population: Those participants with data at six weeks
Measure: Number; unit: percentage of participants
Arm/Group | Oral Iron | IV Iron
Number analyzed (Participants) | 45 | 47
percentage of participants | 75 | 68
Statistical Analysis 1: Comparison: Oral Iron vs IV Iron; Test type: Superiority; p = 0.55, Chi-squared

3. Secondary Outcome: Number of Participants With Adverse Events Judged Related or Possibly Related to Treatment.
Description: Patient reported gastrointestinal or constitutional adverse events
Time Frame: Up to six weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Iron | IV Iron
Number analyzed (Participants) | 46 | 47
Participants | 22 | 11

ADVERSE EVENTS:
Time Frame: Up to six weeks
Arm/Group | Oral Iron | IV Iron
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 22/46 | 11/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Iron (N=46) | IV Iron (N=47)
Constipation (Gastrointestinal disorders) | 8 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 2
Mouth Burn (Gastrointestinal disorders) | 0 | 1 — Occurring at baseline with test dose
Gastric Irritation (Gastrointestinal disorders) | 7 | 5
Arthralgia/myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Edema (General disorders) | 1 | 1
Oral iron intolerance (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-07-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT02499354/Prot_000.pdf
  • Statistical Analysis Plan (2014-07-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT02499354/SAP_001.pdf